CLINICAL TRIAL: NCT07117695
Title: Efficacy of Multidisciplinary Prevention Clinic Model for Cardiovascular Risk Reduction in High Risk Patients
Brief Title: Duke Cardiometabolic Prevention Clinic's Impact on High-risk Cardiovascular Patients With Uncontrolled Risk Factors
Acronym: DUKE PREVENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Barnhill Family Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00109610
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: ASCVD; Hyperlipidemia; Hypertension
Keywords: ASCVD; Cardiometabolic Clinic; Prevention; Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Referral to Cardiometabolic Prevention Clinic (Experimental): Participants referred to the Duke Cardiometabolic Prevention Clinic will be evaluated by a cardiology provider and receive coordinated care based on their risk factors. This may include referrals to specialists in endocrinology, nephrology, or hepatology. A multidisciplinary team will manage their care to help improve heart and metabolic health.
  Interventions: Other: Referral to the Duke Cardiometabolic Prevention Clinic
- Standard of Care Group (No Intervention): Participants in the standard care group will not be contacted directly and will continue their usual care with their primary care provider.

INTERVENTIONS:
Other: Referral to the Duke Cardiometabolic Prevention Clinic — Patients who are referred to the cardiometabolic prevention clinic within the intervention arm will be evaluated first by a cardiology provider (as each patient has a history of ASCVD). On this initial visit, the cardiology provider will assess the patient's risk factor profile - to identify the presence of co-morbid conditions or uncontrolled risk factors. The need for additional referrals to other clinicians within the cardiometabolic clinic will specifically outlined criteria. These referrals will be offered to the patient and facilitated after the first visit. Preventive care will follow routine, evidence-based care. Clinicians within the cardiometabolic prevention clinic will meet bi-weekly to discuss enrolled patients, thus every individual in the intervention arm will receive coordinated, multi-specialty care.
  Arms: Referral to Cardiometabolic Prevention Clinic

SUMMARY:
This project is studying whether a team-based specialty clinic can help people with type 2 diabetes and heart disease better manage their blood pressure and cholesterol. The clinic includes coordinated care from heart doctors, kidney doctors, diabetes specialists, and liver doctors.

The study will compare two groups of patients: one receiving usual care from their primary care provider, and one referred to the Duke Cardiometabolic Prevention Clinic for multidisciplinary care. The main goals are to find out if this clinic improves blood pressure and cholesterol control over 12 months, increases use of recommended heart medications, and reduces hospital visits and other healthcare use.

Participants will be randomly assigned to one of the two groups. Those referred to the clinic will: 1) Meet with a cardiologist for an initial evaluation. 2) Be referred to other specialists (such as endocrinology, nephrology, or hepatology) based on their needs. 3) Receive ongoing, coordinated care from a team of specialists working together to improve their heart and metabolic health.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age
2. Prior history of cardiovascular disease (prior history of CAD, MI, ischemic stroke, PVD, any arterial revascularization)
3. Type 2 Diabetes
4. Uncontrolled sBP AND LDL-C within the preceding 3 months:

   * SBP > 150mmHg on at least 1 occasion in last 3 months, AND
   * LDL > 130mg/dL in last 3 months

     * NOTE: If there are not enough patients with the above inclusion criteria available for enrollment, then we will expand the criteria to include patients with uncontrolled sBP and LDL-C within the last 6 months.

Exclusion Criteria:

1. Currently or previously established with providers in the Duke Cardiometabolic Prevention Clinic (Pagidipati, Shah, McGarrah, Blazing, Kelsey)
2. History of advanced dementia
3. Referred to hospice/on hospice
4. Lives outside of Durham County, Orange County, Wake County, Person County or Granville County
5. End Stage Renal Disease (those on dialysis or with EGFR <20)
6. History of cardiac transplant/Listed for Cardiac Transplant/Followed by Advanced Heart Failure
7. Pregnant/Planning to become pregnant during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-06-02 (Estimated); Primary Completion 2027-09-27 (Estimated); Study Completion 2027-12-27 (Estimated)

PRIMARY OUTCOMES:
Change in LDL-C | Baseline, 12 months after enrollment
  Change in low-density-lipoprotein cholesterol from baseline
Change in Systolic Blood Pressure | Baseline, 12 months after enrollment
  Change in systolic blood pressure from baseline

SECONDARY OUTCOMES:
Number of participants meeting Risk Factor Targets | 12 months after enrollment
  Those achieving both of the following, and of attaining each component individually: systolic blood pressure (sBP) < 130 and low-density-lipoprotein (LDL) < 70mg/dL
Change in Number of participants on Evidence-Based Medication Targets | Baseline, 12 months after enrollment
  Evidence-based medications include (where appropriate) ACE/ARB/ARNI, high-intensity statin, SGLT2i or GLP-1 RA.

OTHER OUTCOMES:
Time to first composite event of all-cause mortality, myocardial infarction, stroke, or coronary revascularization | 12 months after enrollment
Healthcare Utilization: Outpatient Encounters | 12 months after enrollment
  Number of outpatient encounters
Healthcare Utilization: All-cause hospitalizations | 12 months after enrollment
  Number of all-cause hospitalizations
Healthcare Utilization: Number of cardiovascular (CV) hospitalizations | 12 months after enrollment
  CV hospitalizations include those for MI (myocardial infarction), HF (heart failure), stroke, coronary or peripheral revascularization/amputation.

CONTACTS AND LOCATIONS:
Overall Officials: Neha J Pagidipati, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No